CLINICAL TRIAL: NCT06029231
Title: Quantifying Radiation-Induced Skin Reactions: Establishing the Foundation for Future Prediction Models
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chin-Nan Chu, Attending physician, China Medical University Hospital
Other Study IDs: CMUH112-REC1-120
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: radiation-irritated skin; Radiation therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer has the highest incidence rate among female cancers, and breast radiotherapy plays an essential role in the treatment of breast cancer. However, the acute and chronic skin reactions caused by radiotherapy, especially radiation dermatitis, have a significant impact on the physical and mental health of breast cancer patients. Severe acute radiation dermatitis can affect the patient's quality of life and may even lead to treatment interruption, thereby affecting treatment efficacy. Chronic radiation dermatitis can lead to irreversible skin problems, such as "radiation-irritated skin" and skin pigmentation, which can affect the quality of life of breast cancer patients after treatment.

This study aimed to evaluate and examine the skin reactions of 30 breast cancer patients who underwent whole-breast radiotherapy after breast conserving surgery. The subjects returned to the hospital for evaluation every week during radiotherapy, and in the second and sixth weeks after the end of the treatment, they received physical examinations and surveys, including questionnaire surveys, skin observations and measurements. The study lasted for 3 months. Skin observation items included physiological parameters such as skin moisture, temperature, melanin, transepidermal water loss (TEWL), and clinical evaluation of skin reactions by physicians. Through statistical analysis of skin physiological parameters, scientific instruments can quantify the radiation skin reactions traditionally judged by clinical physicians by visual examination and can perform real-time clinical prediction monitoring, which can be used to establish a skin reaction prediction model in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be males or non-pregnant females at least 18 years of age.
* Diagnosis of non-inflammatory breast adenocarcinoma or in situ breast cancer which will be treated by radiotherapy after operation.
* Patient had unilateral breast conservation surgery with or without adjuvant or neoadjuvant chemotherapy or hormonal treatment.
* Patients were scheduled to receive at least five sessions of radiotherapy per week (1 session per day) for at least four weeks using standard irradiation fraction (with at least 1.8 Gy per session) for total dose of at least 45 Gy.
* Participant must give informed consent.

Exclusion Criteria:

* Bilateral breast cancer
* Previous radiotherapy to the chest
* Prior breast reconstructions, implants, and/or expanders
* Known radiosensitivity syndromes (e.g. Ataxia-telangiectasia)
* Collagen vascular disease, vasculitis, unhealed surgical sites, breast infections or systemic lupus erythematosus (SLE)
* Participation in any clinical trial in the prior 30 days from baseline.
* Any condition that, in the judgement of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of non-inflammatory breast adenocarcinoma or in situ breast cancer which will be treated by radiotherapy after operation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
The worst skin toxicity according to CTCAE grading. | 1-Week (Day0), 2-Week (Day7), 3-Week (Day14), 4-Week (Day21), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later
  The worst skin toxicity during radiotherapy and 2 weeks after according to CTCAE grading.

SECONDARY OUTCOMES:
To compare the skin moisture percentage. | 1-Week (Day0), 3-Week (Day14), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  To compare the skin moisture percentage at the radiotherapy site and normal site from baseline to follow-up visit.
To compare the skin trans-epidermal water loss. | 1-Week (Day0), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  To compare the skin trans-epidermal water loss at the radiotherapy site and normal site from baseline to follow-up visit.
To compare the skin temperature of target region. | 1-Week (Day0), 3-Week (Day14), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  To compare the skin temperature of target region at the radiotherapy site and normal site from baseline to follow-up visit.
The score of quality of life with the Skindex-16 questionnaire performed every two weeks. | 1-Week (Day0), 3-Week (Day14), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  The score of quality of life with the Skindex-16 questionnaire performed every two weeks.
Median time to G2 radiation dermatitis development | 1-Week (Day0), 2-Week (Day7), 3-Week (Day14), 4-Week (Day21), 5-Week (Day28), 6-Week (Day35), Post-radiotherapy 2 Week later, Post-radiotherapy 6 Week later
  Median time to G2 radiation dermatitis development

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan